CLINICAL TRIAL: NCT05533125
Title: Rituximab Effect on Decreasing glUcoCorticoid Exposition in PolyMyalgia Rheumatica
Brief Title: Rituximab Effect on Decreasing glUcoCorticoid Exposition in PolyMyalgia Rheumatica Patients Recently Diagnosed
Acronym: REDUCE-PMR-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: Dutch Arthritis Association (Industry); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDUCE PMR 1
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): 1000mg rituximab intravenously once
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): 0mg rituximab (placebo) intravenously once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000mg in 250ml NaCl 0.9% intravenously with usual premedication
  Other Names: Rixathon; MabThera; Ruxience; Truxima
  Arms: Rituximab
Drug: Placebo — Placebo in 250ml NaCl 0.9% intravenously with usual premedication
  Arms: Placebo

SUMMARY:
Polymyalgia rheumatica (PMR) is prevalent among elderly. Untreated, it leads to major reduction in quality of life. Glucocorticoids are the cornerstone of treatment, but have drawbacks, warranting glucocorticoid sparing treatment. A proof of concept study on Rituximab (RTX) vs placebo showed efficacy in 48 vs 21%(p=0.049) in glucocorticoid free remission after 21 weeks (Marsman et al. 2021). Though promising, the short study duration and small sample size require further confirmation. Therefore a larger randomised controlled trial with longer follow up will be performed on RTX efficacy on glucocorticoid free remission in newly diagnosed PMR patients during glucocorticoid taper.

ELIGIBILITY:
Inclusion Criteria:

* Polymyalgia rheumatica diagnosis fulfilling the 2012 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria
* Diagnoses less than 12 weeks ago
* Glucocorticoid treatment less than 8 weeks and with dose equivalent of prednisolone ≤ 30 mg/day
* Informed consent

Exclusion Criteria:

* treatment with systemic immunosuppressants (other than glucocorticoids) 3 months prior to inclusion;
* (clinical) suspect concomitant giant cell arteritis or other rheumatic inflammatory diseases;
* concomitant conditions that might significantly interfere with PMR pain or movement evaluation as judged by the investigator;
* previous hypersensitivity for RTX or contra-indications to RTX.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Between group difference in percentage of patients in glucocorticoid-free remission | At week 52
  Between group difference in percentage of patients in glucocorticoid-free remission (PMR activity score < 10) at week 52

SECONDARY OUTCOMES:
Percentage of patients in glucocorticoid-free remission | 21 weeks
  Percentage of patients in glucocorticoid-free remission
Percentage of patients with glucocorticoid dose of ≤5mg/day | 52 weeks
  Percentage of patients with glucocorticoid dose of ≤5mg/day
Number of relapses | 52 weeks
  Number of relapses
Time to glucocorticoid-free remission | 52 weeks
  Time to glucocorticoid-free remission in days during the study period
Time to relapse | 52 weeks
  Time to relapse in days during the study period
Cumulative glucocorticoid dose | 52 weeks
  Cumulative glucocorticoid dose
Percentage of patients needing RTX/Placebo retreatment | 52 weeks
  Percentage of patients needing RTX/Placebo retreatment
Adverse events | 52 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Aatke van der Maas, MD PhD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartensklineik, Ubbergen, Gelderland, Netherlands

REFERENCES:
- [Derived] Sun MM, Pope JE. Polymyalgia rheumatica and giant cell arteritis: diagnosis and management. Curr Opin Rheumatol. 2025 Jan 1;37(1):32-38. doi: 10.1097/BOR.0000000000001059. Epub 2024 Oct 14. PMID 39400109